CLINICAL TRIAL: NCT02453347
Title: Cranial Electrotherapy Stimulation (CES) Therapy for PTSD and Anxiety in OEF/OIF Veterans With Mild TBI
Brief Title: Cranial Electrotherapy Stimulation (CES) Therapy
Acronym: CES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-352H (UTHSCSA IRB)
Record Dates: First submitted 2015-05-14; First posted 2015-05-25 (Estimated); Results first posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2017-11

CONDITIONS: TBI; Anxiety; PTSD; Depression
Keywords: Stable chronic medical conditions; No current alcohol or substance abuse; Alpha Stim
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic; Depression; Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CES Therapy (Experimental): All participants will complete CES treatment over the course of four weeks. Assessments will take place at baseline and at post-test four weeks later.
  Interventions: Device: CES Therapy

INTERVENTIONS:
Device: CES Therapy — Cranial Electrotherapy Stimulation (CES) may serve as an effective complimentary, noninvasive/non-pharmacological treatment for this Veteran population. CES is administered through a therapeutic device (such as Alpha-Stim®) marketed and approved by the FDA to treat insomnia, depression, anxiety, and pain.
  Other Names: Cranial Electrotherapy Stimulation (CES) Therapy; Alpha Stim

SUMMARY:
The primary aim of this proposed study is to gather preliminary data for CES use in treating PTSD and anxiety symptoms in OEF/OIF Veterans with PTSD and a history of TBI.

DETAILED DESCRIPTION:
Veterans from conflicts in Afghanistan and Iraq exhibit numerous signature injuries to include posttraumatic stress disorder (PTSD), traumatic brain injury (TBI), and anxiety. These three conditions commonly co-occur together, which presents treatment challenges. First, current treatment guidelines focus on treating each of these conditions individually and do not sufficiently account for comorbid presentation. As a consequence, Veterans with comorbid disorders may have poor clinical health outcomes despite receiving treatment. Second, treating anxiety among Veterans with comorbid PTSD and TBI involves medications that may have limited efficacy (e.g., PTSD medications) or side effects (e.g., drug interactions or diminished cognitive function).

Given these treatment challenges, Cranial Electrotherapy Stimulation (CES) may serve as an effective complimentary, noninvasive/non-pharmacological treatment for this Veteran population. Briefly, CES is administered through a therapeutic device (such as Alpha-Stim®) marketed and approved by the FDA to treat insomnia, depression, anxiety, and pain. Additionally, both the Department of Defense (DoD) and Veterans Health Affairs (VHA) prescribe CES to treat trauma-related conditions. CES treatment involves transcutaneous application of pulsed micro-currents of <1000 μA to the patient's head and these currents are tailored specifically for each patient. The studies that have examined efficacy for CES therapy in treating anxiety have shown some positive effects, however, the patient populations were typically small, sometimes limited to case reports, and outcome measures varied significantly. A meta-analysis performed on CES studies over two decades ago found evidence for CES treatment over sham groups, but most of the studies reviewed were missing data and study personnel were not always blinded to the groups. Additionally, CES has showed a significant improvement in anxiety symptoms after of CES therapy in 12 adult patients diagnosed with generalized anxiety disorder (GAD; Bystritsky et al., [2008]). The success of CES in treating anxiety may indicate a suitable signal for exploring its use in PTSD samples (Novakovic et al. [2011]). Given the relatively few CES studies available in the scholarly literature, a 2009 Cochrane Systematic Review found insufficient evidence to support using CES to manage persistent TBI symptoms. While some of these studies are encouraging, the device has not been clearly demonstrated to be effective in the multi-morbid OEF/OIF/OND Veteran population. Additionally, little information is known about the mechanism of action for CES.

ELIGIBILITY:
Inclusion Criteria:

* Male outpatient, OEF/OIF/OND Veterans diagnosed during the course of clinical care with mild TBI and PTSD, and screened positive for anxiety
* Good medical health and stable chronic medical conditions.
* No current alcohol or substance abuse.

Exclusion Criteria:

* Patients with moderate or severe TBI or seizure disorders.
* Prior CES use
* Diagnosis of Bipolar Disorder, Schizophrenia, or other psychiatric condition that would require inpatient hospitalization or medical disease that would impair reliable participation in the trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Jaramillo, M.D., Ph.D., Principal Investigator — San Antonio Polytrauma Center South Texas Veterans Health Care System
Locations (1):
- Audie L. Murphy VA Hospital, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CES Therapy
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CES Therapy
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (8.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Region from which participants are enrolled
  participants
    United States | 6

OUTCOME MEASURES:

1. Primary Outcome: PCL-5 (Post Traumatic Stress Disorder Checklist for the Diagnostic and Statistical Manual of Mental Disorders) for Use in Treating PTSD Symptoms
Description: To measure the effect of Cranial Electrotherapy Stimulation (CES) use on symptoms related to PTSD.
  The PCL-5 is a self-report measure that can be completed by patients in a waiting room prior to a session or by participants as part of a research study.
  The survey has 20 questions scored as:
  0=Not at all
  1. A little bit
  2. Moderately
  3. Quite a bit
  4. Extremely Interpretation of the PCL-5 should be made by a clinician. The total symptom severity score is obtained by summing the scores for each of the 20 items and ranges from 0 to 80. The lower the score, the less severe the symptoms of PTSD, the higher the score, the more severe the symptoms. For a person to have a probable diagnosis of PTSD sufficient criteria must be moderately to extremely met in each of the four symptom groups (i.e., one or more of questions 1-5, either question 6 or 7, two or more of questions 8-14, two or more of questions 15-20). In addition, a score of 38 or higher indicates probable PTSD in veterans.
Time Frame: Four Weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CES Therapy
Number analyzed (Participants) | 6
scores on a scale | 44.25 (17.87)

2. Primary Outcome: State-Trait Anxiety Inventory (STAI)
Description: To measure the effect of CES use on trait and state anxiety. These scales comprise 20 items each and are scored on 4-point forced-choice response scales from 1 (seldom) to 4 (frequent). Scores range from 20 to 80, with higher scores suggesting greater levels of anxiety.The state and trait anxiety scales both range from 20 to 80 and are combined to yield a total score ranging from 40 to 160, where low scores suggest mild anxiety, median scores suggest moderate anxiety, and high scores suggest severe anxiety. Both scales include direct (presence of anxiety) and reverse-worded (absence of anxiety) items. Reverse-worded item scores are reverse scored and then totaled with the remaining items.
Time Frame: Four Weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CES Therapy
Number analyzed (Participants) | 6
scores on a scale | 81.375 (16.85)

3. Primary Outcome: Beck Depression Inventory (BDI)
Description: A 21 question set to assess subjects feelings in the last week. Each question has a set of at least 4 possible responses, ranging in intensity:
  (0) I do not feel sad.
  1. I feel sad.
  2. I am sad all the time and I can't snap out of it.
  3. I am so sad or unhappy that I can't stand it. When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score ranging from 0 to 63 is compared to a key to determine the depression's severity. Higher total scores indicate more severe depressive symptoms.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score
Arm/Group | CES Therapy
Number analyzed (Participants) | 6
score | 25 (13.9)

4. Primary Outcome: TFI (Tinnitus Functional Index)
Description: To measure the severity of tinnitus. The survey consists of 25 questions ranked from 0 (did not interfere) to 10 (completely interfered). At least 19 of the 25 questions are required to be answered, and rankings are added together to give a maximum possible score of 250, which would be the most severe interference by tinnitus.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CES Therapy
Number analyzed (Participants) | 6
scores on a scale | 94.875 (45.26)

5. Primary Outcome: MPAI (Mayo Portland Adaptability Inventory)
Description: The inventory consists of 29 items in 3 subscales (Ability, the Adjustment and Participation Index) plus an additional 6 items that are not included in the MPAI-4 score. The first 29 scale items are intended to reflect the current status of the individual with brain injury without attempting to determine whether their status might be influenced by factors other than ABI (acquired brain injury). Items are scored from 0 to 4, with 0 being the most favorable score for each item, with a cumulative score ranging from 0 to 116 for all the items. A lower score indicates better adaptability.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CES Therapy
Number analyzed (Participants) | 6
scores on a scale | 48 (16.34)

6. Primary Outcome: WAIS (Wechsler Adult Intelligence Scale) Symbol Search
Description: The Symbol Search subtest of the Wechsler Adult Intelligence scale designed to assess information processing speed and visual perception with a minimum score of 0 as the lowest (worst performance) to 60 as the highest score (best performance).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CES Therapy
Number analyzed (Participants) | 6
scores on a scale | 26.75 (10.41)

7. Primary Outcome: WAIS Coding - Wechsler Adult Intelligence Scale
Description: The test has two batteries of subtests grouped into two general areas: 1) Verbal scales; and 2) Performance scales. The Verbal scales measure general knowledge, language, reasoning, and memory skills, while the Performance scales measure spatial, sequencing, and problem-solving skills.
  The tests are administered to individual examinees by trained examiners, using a complex set of test materials. Testing requires approximately 90 minutes. Raw scores on each test are converted to standard scores with a mean of 10 and a standard deviation of 3. Scale scores in the Verbal battery are summed and converted to a Verbal Intelligence Quotient (IQ) score; the same is done for the Performance scale scores which yield the Performance IQ score. In turn, the Verbal and Performance IQ scores are summed and converted to obtain the Full Scale (overall) IQ score with a mean of 100 and a standard deviation of 15. Higher scores indicate a higher IQ.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CES Therapy
Number analyzed (Participants) | 6
scores on a scale | 55.5 (23.9)

8. Secondary Outcome: Dizziness- NSI (Neurobehavioral Symptom Inventory)
Description: To measure the effect of CES use on somatic symptoms related to TBI (Traumatic Brain Injury), including dizziness. The assessment scale rate 22 symptoms that may have disturbed subjects from 0 = no symptoms to 4 = very severe in the previous 2 weeks. The scores are summed to yield a total score ranging from 0 to 88, where the higher the point value, the greater the symptoms.
Time Frame: Four Weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CES Therapy
Number analyzed (Participants) | 6
scores on a scale | 40.8 (21.5)

9. Secondary Outcome: Headache - HIT6 (Headache Impact Test)
Description: To assess for improvements in measures of somatic symptoms related to TBI (headaches). The test is scored by adding points to 6 different categories related to frequency and severity of symptoms. The 6 category scores are summed to yield a total score ranging from 36 to 78. Fewer points signify less severity and higher point scores signify more severe symptoms according to patient assessment.
Time Frame: Four Weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CES Therapy
Number analyzed (Participants) | 6
scores on a scale | 62.37 (5.5)

10. Secondary Outcome: Sleep - Pittsburgh Sleep Quality Index (PSQI)
Description: To assess for improvements in measures of somatic symptoms related to TBI (insomnia). The scoring consists of 19 items, the PSQI measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction.
  Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Time Frame: Four Weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CES Therapy
Number analyzed (Participants) | 6
scores on a scale | 10.5 (5.26)

ADVERSE EVENTS:
Time Frame: From baseline to 12 months
Arm/Group | CES Therapy
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No